CLINICAL TRIAL: NCT00477217
Title: A Randomized, Double-blind, Placebo-controlled, Proof of Concept Study of Zoledronic Acid in Spontaneous Osteonecrosis of the Knee (SONK)
Brief Title: Zoledronic Acid Treatment of Spontaneous Osteonecrosis of the Knee
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HAU21
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Osteonecrosis
Keywords: Osteonecrosis; zoledronic acid; knee
MeSH Terms: conditions — Osteonecrosis | interventions — Zoledronic Acid

ARMS (1):
- 1 (Other)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: Reclast, Aclasta

SUMMARY:
This study will assess the safety and efficacy of zoledronic acid in patients presenting with spontaneous osteonecrosis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40-85 years of age
* Diagnosis of painful osteonecrosis of the knee within the last month.

Exclusion Criteria:

* Intravenous (iv) bisphosphonates within the last 2 years.
* Abnormal thyroid, kidney or liver function.
* Abnormal blood calcium or alkaline phosphatase levels.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline after 3 months in a) knee pain scores (using the KOOS pain subscale), and b) volume of osteonecrotic lesion (indicated by bone marrow oedema) on MRI. | 3 months

SECONDARY OUTCOMES:
Changes from baseline after 6 months in a) knee pain scores (using the KOOS pain subscale), and b) volume of osteonecrotic lesion (indicated by bone marrow oedema) on MRI. | 6 months
Safety as assessed by adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis ., Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Gordon, Australia